CLINICAL TRIAL: NCT05909397
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL, MULTICENTER STUDY OF VEPDEGESTRANT (ARV-471/PF-07850327) PLUS PALBOCICLIB VERSUS LETROZOLE PLUS PALBOCICLIB FOR THE TREATMENT OF PARTICIPANTS WITH ESTROGEN RECEPTOR POSITIVE, HER2 NEGATIVE BREAST CANCER WHO HAVE NOT RECEIVED ANY PRIOR SYSTEMIC ANTI CANCER TREATMENT FOR ADVANCED DISEASE (VERITAC-3)
Brief Title: Vepdegestrant (ARV-471/PF-07850327) + Palbociclib vs Letrozole + Palbociclib in ER(+)/HER2(-) Advanced Breast Cancer
Acronym: VERITAC-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4891002; 2022-500545-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Advanced tumor of the breast; Advanced cancer of the breast; Breast neoplasm; Breast tumor; Breast cancer; ER positive; Estrogen receptor positive; HER2-negative; Metastatic breast cancer; Palbociclib; Letrozole; ARV-471; Vepdegestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Investigational Arm) (Experimental): Participants will receive:
  * Vepdegestrant, orally, once daily, continuously, in a 28-day cycle, plus
  * Palbociclib, orally, once daily for 21 consecutive days followed by 7 days off treatment in a 28 day cycle
  Interventions: Drug: Vepdegestrant (ARV-471/PF-07850327); Combination Product: Palbociclib
- Arm B (Comparator Arm): (Active Comparator): Participants will receive:
  * Letrozole, orally, once daily, continuously, in a 28-day cycle, plus
  * Palbociclib, orally, once daily for 21 consecutive days followed by 7 days off treatment, in a 28-day cycle.
  Interventions: Drug: Letrozole; Combination Product: Palbociclib

INTERVENTIONS:
Drug: Vepdegestrant (ARV-471/PF-07850327) — Pharmaceutical form: Tablets. Route of Administration: Oral
  Other Names: Vepdegestrant
  Arms: Arm A (Investigational Arm)
Combination Product: Palbociclib — Pharmaceutical form: Capsules. Route of Administration: Oral.
  Other Names: IBRANCE®
  Arms: Arm A (Investigational Arm)
Drug: Letrozole — Pharmaceutical form: Capsules. Route of Administration: Orally
  Other Names: FEMARA®
  Arms: Arm B (Comparator Arm):
Combination Product: Palbociclib — Pharmaceutical form: Capsules. Route of Administration: Oral.
  Other Names: IBRANCE®
  Arms: Arm B (Comparator Arm):

SUMMARY:
The purpose of this study is to understand the safety and effects of the study medicine vepdegestrant (ARV-471/PF-07850327) given together with palbociclib in advanced breast cancer. In particular, the study will compare the combination of vepdegestrant plus palbociclib to standard of care therapy (letrozole plus palbociclib). Both letrozole and palbociclib are medicines already used for treatment of breast cancer. Vepdegestrant is a new medicine under study.

This study is seeking participants who have breast cancer that:

* Have a locally advanced or metastatic disease and cannot be fully cured by surgery or radiation therapy. A metastatic disease is when disease has spread to other parts of the body.
* Is sensitive to hormonal therapy such as tamoxifen. This is called estrogen receptor positive disease.
* Have not received any prior medicine for advanced disease. Example medications include tamoxifen or letrozole or exemestane.

The study will have an open-label SLI (study lead-in) before initiation of Phase 3 trial. During SLI, two dose levels of palbociclib in combination with vepdegestrant will be explored in parallel. Assignment to the palbociclib dose is by chance. Half of the participant will receive one dose and the other half another palbociclib dose. The purpose of SLI is to determine the recommended Phase 3 dose of palbociclib to be administered in combination with vepdegestrant.

In the Phase 3, half of the participants will take vepdegestrant plus palbociclib while the other half will take letrozole plus palbociclib. In both SLI and Phase 3, participants will take the study medicines by mouth, with food, once a day. Participants will take the study medicines until breast cancer increase in size or side effects become too severe. Side effects refer to unwanted reactions to medications. Participants will visit the study clinic about once every 4 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that vepdegestrant (ARV-471) in combination with palbociclib provides superior clinical benefit compared to letrozole in combination with palbociclib in participants with ER(+)/HER2(-) aBC who have not received any prior systemic anti-cancer therapies for their locoregionally advanced or metastatic disease.

The study will have a Study Lead-in (SLI) and a Phase 3. In the SLI, 50 participants (approximately 25 each arm) will be randomly assigned on a 1:1 basis to one of the two dose levels (DLs). In the randomized Phase 3, approximately 1130 eligible participants (approximately 565 each arm) will be randomized in a 1:1 ratio to the Experimental Arm (ie, vepdegestrant plus palbociclib at RP3D determined in the SLI) or Control Arm (ie, letrozole plus palbociclib at the registered doses). Randomization will be stratified by menopausal status at study entry, visceral disease and de novo metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with loco-regional recurrent or metastatic disease not amenable to curative treatment
* Confirmed diagnosis of ER+/HER2- breast cancer
* No prior systemic treatment for loco-regional recurrent or metastatic disease
* Measurable disease evaluable per Response Evaluation Criterion in Solid Tumors (RECIST) v.1.1 or non-measurable bone-only disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Phase 3 only: Participants should be willing to provide blood and tumor tissue

Exclusion Criteria:

* Disease recurrence while on, or within 12 months of completion of adjuvant endocrine therapy
* Prior treatment with cyclin dependent kinase 4/6 inhibitors (CDK4/6i), vepdegestrant, fulvestrant, elacestrant and other investigational drugs including novel endocrine therapies, any selective estrogen receptor degraders (SERDs), covalent antagonists (SERCAs) and complete ER antagonists (CERANs).
* Inadequate liver, kidney and bone marrow function
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Refractory nausea and vomiting, inability to swallow capsules and tablets whole, chronic gastrointestinal diseases, significant gastric (total or partial) or bowel resection that would preclude adequate absorption of study interventions.
* Current use or anticipated need for food, herbal supplements or drugs that are known strong CYP3A4 inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Study Lead-in (SLI): Incidence of Grade 4 neutropenia | From randomization date up to Cycle 4 (each cycle is 28 days).
  It is defined as the number of participants with Grade 4 neutropenia AE (graded by NCI CTCAE v.5.0) with onset within the first 4 cycles divided by the number of participants.
SLI: Incidence of dose reduction | From randomization date up to Cycle 4 (each cycle is 28 days).
  It is defined as the number of participants reducing the dose of palbociclib and/or vepdegestrant due to any cause occurring within the first 4 cycles divided by the number of participants.
SLI: Incidence of drug discontinuation. | From randomization date up to Cycle 4 (each cycle is 28 days).
  It is defined as the number of participants discontinuing palbociclib and/or vepdegestrant due to any cause occurring within the first 4 cycles divided by the number of participants.
Phase 3: Progression-Free Survival | From randomization date, every 12 weeks, to date of first documentation of progression or death, up to approximately 4 years.
  Progression-free survival is defined as the time interval from the date of randomization to the date of first documented tumor progression determined by Blinded Independent Central Review (BICR) as per Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) or death due to any cause, whichever come first.

SECONDARY OUTCOMES:
SLI and Phase 3. Objective Response Rate | From randomization date, every 12 weeks, to the date of progression or death (up to approximately 4 years).
  Objective response rate is defined as the proportion of participants who have a confirmed CR or PR, as best overall response determined by Investigators (SLI) or by BICR (Phase 3) as per RECIST version 1.1, from the date of randomization to the date of disease progression or death due to any cause, whichever occurs first.
SLI and Phase 3: Duration of Response | From the date of the first objective response, every 12 weeks, to the date of disease progression or death (up to approximately 4 years).
  Duration of response is defined as the time from first documented evidence of CR or PR until progressive disease (PD) determined by Investigators (SLI) or by BICR (Phase 3) as per RECIST version 1.1 or death due to any cause, whichever occurs first.
SLI and Phase 3: Clinical Benefit Rate | Every 12 weeks From randomization date, every 12 week, to the date of progression or death (up to approximately 4 years).
  Clinical benefit rate is defined as the proportion of participants who have a confirmed CR, PR at any time or SD or non CR/non PD for at least 24 weeks determined by Investigators (SLI) or by BICR (Phase 3) as per RECIST version 1.1, from the date of randomization until disease progression or death due to any cause, whichever occurs first.
Phase 3: Overall Survival | From randomization date, every 3 months, to date of death (up to approximately 6 years)
  Overall survival is defined as the time interval from the date of randomization to the date of documented death, due to any cause.
SLI and Phase 3: Incidence of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From baseline to date to end of treatment (up to approximately 4 years)
  It is defined as the number of participants with TEAEs and SAEs divided by the number of participants. AEs and SAEs will be graded according to NCI CTCAE V5.0.
SLI and Phase 3: Incidence of laboratory abnormalities | From baseline to end of treatment (up to approximately 4 years)
  It is defined as the number of participants with laboratory abnormalities divided by the number of participants. Laboratory abnormalities will be graded according to NCI CTCAE V5.0.
SLI and Phase 3: Incidence of Electrocardiogram (ECG) Abnormalities | From baseline up to the end of treatment (up to approximately 4 years)
  It is defined as the number of participants with ECG abnormalities divided by the number of participants. ECG abnormalities will be graded according to NCI CTCAE V5.0.
SLI and Phase 3: Plasma concentrations of vepdegestrant and palbociclib | From randomization date up to Cycle 5 (each cycle is 28 days)
  Plasma concentrations of vepdegestrant and palbociclib
Phase 3: Health state utility and health status will be assessed using the European Quality of Life Group questionnaire with 5 dimensions and 5 levels per dimension (EQ-5D-5L) | From baseline, each cycle up to cycle 3, then every odd cycle to end of treatment (up to approximately 4 years). Each cycle is 28 days
  Change from baseline between treatment comparison in Quality of Life using the EQ-5D 5L questionnaire.
Phase 3: Disease-related Quality of Life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ-C30) | From baseline, each cycle up to Cycle 3, then every odd cycle to end of treatment (up to approximately 4 years). Each cycle is 28 days.
  Change from baseline between treatment comparison in Quality of Life using the EORTC QLQ-C30 questionnaire.
Phase 3: Disease- and treatment-related Quality of Life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) breast cancer module (QLQ-BR23) questionnaire. | From baseline, each cycle up to Cycle 3, then every odd cycle to end of treatment (up to approximately 4 years). Each cycle is 28 days.
  Change from baseline between treatment comparison in Quality of Life Using the EORTC QLQ-BR23 (Breast) questionnaire.
Phase 3: Changes from baseline in plasma ctDNA (Circulating Deoxyribonucleic Acid) | From baseline to end of treatment (up to approximately 4 years)
  Quantitative changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (3):
  - BRCR Global, Plantation, Florida
  - BRCR Medical Center Inc, Plantation, Florida
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (2):
  - Cancer Research SA, Adelaide, South Australia
  - Barwon Health, Geelong, Victoria
- Brazil (4):
  - Hospital Santa Rita de Cassia, Vitória, Espírito Santo
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
- China (4):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Italy (3):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
- Japan (3):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Slovakia (2):
  - Nemocnica na okraji mesta n o, Partizánske
  - Fakultna nemocnica s poliklinikou J.A. Reimana Presov, Prešov
- Spain (6):
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [barcelona]
  - Hospital Universitari Dexeus, Barcelona, Catalunya [cataluña]
  - Complejo Hospitalario de Jaén, Jaén, JAÉN
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Unviersitario Virgen Nieves, Granada
  - Hospital Clinico San Carlos, Madrid
- Tumor Zentrum Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891002